CLINICAL TRIAL: NCT04342325
Title: Open-label, Multiple-center, Dose-Escalation Study to Evaluate the Safety and Tolerability of ADR-001 for the Treatment for Immunoglobulin A (IgA) Nephropathy
Brief Title: The Clinical Trial of ADR-001 for IgA Nephropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nagoya University (Other)
Collaborators: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shoichi Maruyama MD PhD, Professor at Department of Nephrogy, Graduate school of Medicine, Nagoya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMCR013; jRCT2043200002 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Glomerulonephritis , IGA
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADR-001 (Experimental): Intravenous infusion of ADR-001 (Mesenchymal stem cell)
  Interventions: Biological: infusion of ADR-001 (Mesenchymal stem cell)

INTERVENTIONS:
Biological: infusion of ADR-001 (Mesenchymal stem cell) — Once or twice with two week interval at a dose of 100 x 10 ^ 6 cells.

SUMMARY:
The purpose of this study is to evaluate the safety and the tolerability of ADR-001 in Immunoglobulin A (IgA) Nephropathy patients. In addition, the investigators will evaluate the efficacy of ADR-001 for IgA Nephropathy patients.

ELIGIBILITY:
Inclusion Criteria:

1. IgA nephropathy diagnosed by renal biopsy.
2. Meet any of the following criteria.

   i. Urinary protein at screening is 0.5 g / gCr or more and eGFR is 60 mL / min / 1.73m^2 or more even if corticosteroids are used for 6 months or more before screening.

   ii. Urine protein of 1.0 g / gCr or more and eGFR of 30 mL / min / 1.73 m^2 or more and less than 60 mL / min / 1.73 m^2 at screening even if corticosteroids are used for 6 months or more before screening.

   iii. Urine protein of 0.5 g / gCr or more and less than 1.0 g / gCr at screening and eGFR of 20 mL / min / 1.73m^2 or more and 60 mL / min / 1.73m^2 or urine protein of 1.0 g / gCr or more at screening And eGFR is 20 mL / min / 1.73m^2 or more and less than 30 mL / min / 1.73m^2.
3. Over 20 years old.
4. Able to provide informed consent.

However, in the first cohort, only 2) -i is applied in the selection criteria 2), and in the second cohort, 2) -i, ii, and iii are applied.

Exclusion Criteria:

1. Nephropathy other than IgA nephropathy, and primary and secondary nephrotic syndrome.
2. Start or increase drug therapy for IgA nephropathy with corticosteroids, immunosuppressants, renin angiotensin system (RAS ) inhibitors, antiplatelet drugs, anticoagulants (warfarin), and n-3 fatty acids (fish oil) within 3 months . Palatal tonsillectomy within 6 months.
3. Treatment with other cells.
4. Participated within 3 months or participating in other clinical trials .
5. Penal transplantation within 3 years or scheduled.
6. Diabetics not well controlled.
7. Malignant neoplasm or history of malignant neoplasm within 5 years, or judged possibility of malignant tumor.
8. Suspected of active infection.
9. Positive for hepatitis B (HB), hepatitis C virus (HCV),human Immunodeficiency virus (HIV), human T-cell leukemia virus 1 (HTLV-1) or syphilis.
10. History of severe hypersensitivity or anaphylactic reaction.
11. Allergic to penicillin antibiotics, aminoglycoside antibiotics or dimethyl sulfoxide (DMSO).
12. Serious complications not related to IgA nephropathy.
13. Bleeding or may bleed, shallow days after surgery or trauma to the central nervous system, history of hypersensitivity to components of heparin preparations, history of heparin-induced thrombocytopenia Previous patient.
14. During pregnancy, lactation, may be pregnant or both men and women who do not agree to give birth control under the guidance of the investigator or investigator during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | until 6 weeks after first administration
  Any adverse events are summarized.

SECONDARY OUTCOMES:
Clinical remission (proteinuria, hematuria) | at 2, 4, 6, 12, 26, 38 and 52 weeks after first administration
  Ratio and time frame to achieve remission are summarized.
Proteinuria | at 2, 4, 6, 12, 26, 38 and 52 weeks after first administration
  Change from baseline value and ratio to achieve threshold are summarized.
Hematuria | at 2, 4, 6, 12, 26, 38 and 52 weeks after first administration
  Change from baseline value and ratio to achieve threshold are summarized.
Estimated glomerular filtration rate (eGFR) | at 2, 4, 6, 12, 26, 38 and 52 weeks after first administration
  Change from baseline value are summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Shoichi Maruyama, MD, PhD, Study Chair — Nagoya University
Locations (2):
- Japan (2):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanaka A, Furuhashi K, Fujieda K, Horinouchi A, Maeda K, Saito S, Mimura T, Saka Y, Naruse T, Ishimoto T, Kato N, Kosugi T, Kinoshita F, Kuwatsuka Y, Nakai Y, Maruyama S. Safety and Tolerability of Adipose-Derived Mesenchymal Stem Cell (ADR-001) Therapy for IgA Nephropathy. Kidney360. 2024 Nov 1;5(11):1692-1705. doi: 10.34067/KID.0000000000000563. Epub 2024 Aug 26. PMID 39186380
- [Derived] Tanaka A, Furuhashi K, Fujieda K, Maeda K, Saito S, Mimura T, Saka Y, Naruse T, Ishimoto T, Kosugi T, Kinoshita F, Kuwatsuka Y, Shimizu S, Nakai Y, Maruyama S. Protocol for a Phase 1, Open-Label, Multiple-Center, Dose-Escalation Study to Evaluate the Safety and Tolerability of ADR-001 in the Treatment of Immunoglobulin A Nephropathy. Front Med (Lausanne). 2022 May 27;9:883168. doi: 10.3389/fmed.2022.883168. eCollection 2022. PMID 35692547